CLINICAL TRIAL: NCT03273413
Title: Statin Therapy in Patients With Early Stage ADPKD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-0678
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: ADPKD; Autosomal Dominant Polycystic Kidney
Keywords: Pravastatin; Statin
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Pravastatin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel study design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive inactive 40 mg tablets of placebo everyday for 6 weeks. If well tolerated, participants will continue taking inactive 40 mg dose of placebo everyday for 2 years.
  Interventions: Drug: Placebo
- Pravastatin (Active Comparator): Participants will receive 40 mg tablets of pravastatin everyday for 6 weeks. If well tolerated, participants will continue taking 40 mg dose of pravastatin everyday for 2 years.
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — Anti-inflammatory, anti-oxidative stress, and anti-proliferative therapy
  Arms: Pravastatin
Drug: Placebo — Inactive tablet
  Arms: Placebo

SUMMARY:
This study plans to learn if pravastatin is helpful in slowing down the progression of kidney disease in adults with autosomal dominant polycystic kidney disease (ADPKD). Pravastatin has been approved by the Food and Drug Administration (FDA) for adults for treatment of hyperlipidemia (high cholesterol levels). The investigators are using pravastatin in this study as an investigational drug for treatment of ADPKD.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial designed to assess the efficacy and benefits of pravastatin therapy in adults with ADPKD by evaluating 1) kidney volume as measured by kidney magnetic resonance imaging (MRI); 2) renal blood flow as measured by kidney magnetic resonance angiography (MRA); 3) kidney function as assessed by Glofil-125; 4) plasma and urine protein markers that will allow a better understanding of how pravastatin works in ADPKD; and 5) blood vessel stiffness as measured by carotid-femoral pulse wave velocity. These parameters will be measured at baseline and after 2 years of pravastatin or placebo treatment in 150 patients with ADPKD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADPKD
* Total kidney volume >500 mL
* Estimated glomerular filtration rate (GFR) ≥60 mL/min/1.73m^2
* Controlled blood pressure <140/80 mmHg

Exclusion Criteria:

* Uncontrolled hypertension
* Diabetes mellitus
* Renal disease, renal cancer, single kidney, recent renal surgery, or acute kidney injury
* Unstable angina
* Coronary artery disease
* Prior ischemic stroke
* Other clinical indication for a statin
* History of hospitalizations within the last 3 months
* Hepatic impairment or liver function abnormalities
* Secondary hypercholesterolemia or hypocholesterolemia
* Use of tolvaptan, gemfibrozil, other fibrates, niacin, clarithromycin, or cyclosporine
* Hypersensitivity to statins
* Immunosuppressive therapy within the last year
* Clinical contraindication for an MRI (i.e. implants, pacemaker, claustrophobia)
* Hypersensitivity to iodine
* Pregnant or breast feeding
* Current tobacco use
* Alcohol abuse or dependence

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Total Kidney Volume | Baseline, 2 years
  Total kidney volume as assessed by renal MRI, at baseline and after 2 years of treatment

SECONDARY OUTCOMES:
Change in Renal Blood Flow | Baseline, 2 years
  Renal blood flow, as assessed by renal MRA, at baseline and after 2 years of treatment
Change in Kidney Function | Baseline, 2 years
  Glomerular filtration rate (GFR), as assessed by Glofil-125, at baseline and after 2 years of treatment
Change in Circulating Inflammatory Markers | Baseline, 2 years
  Plasma levels of inflammatory cytokines and growth factors at baseline and after 2 years of treatment
Change in Circulating Markers of Oxidative Stress | Baseline, 2 years
  Plasma levels of oxidative stress markers at baseline and after 2 years of treatment
Change in Urinary Epithelial Cells | Baseline, 2 years
  Urinary epithelial cell protein expression, as assessed by immunofluorescence, at baseline and after 2 years of treatment

OTHER OUTCOMES:
Change in Blood Vessel Stiffness | Baseline, 2 years
  Blood vessel stiffness, as assessed by carotid-femoral pulse wave velocity, at baseline and after 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michel Chonchol, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver Anschutz Medical Campus, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cadnapaphornchai MA, George DM, McFann K, Wang W, Gitomer B, Strain JD, Schrier RW. Effect of pravastatin on total kidney volume, left ventricular mass index, and microalbuminuria in pediatric autosomal dominant polycystic kidney disease. Clin J Am Soc Nephrol. 2014 May;9(5):889-96. doi: 10.2215/CJN.08350813. Epub 2014 Apr 10. PMID 24721893
- [Derived] Gitomer BY, Ostrow A, Wang W, George D, Coleman E, Nowak KL, Cadnapaphornchai MA, Patel NU, Steele C, Jovanovich A, Klawitter J, Farmer B, You Z, Chonchol M. A randomized controlled trial evaluated the effect of pravastatin on kidney disease outcomes in adult patients with early-stage autosomal dominant polycystic kidney disease. Kidney Int. 2025 Oct 10:S0085-2538(25)00780-X. doi: 10.1016/j.kint.2025.08.037. Online ahead of print. PMID 41077128
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Gitomer BY, Wang W, George D, Coleman E, Nowak KL, Struemph T, Cadnapaphornchai MA, Patel NU, Jovanovich A, Klawitter J, Farmer B, Ostrow A, You Z, Chonchol M. Statin therapy in patients with early-stage autosomal dominant polycystic kidney disease: Design and baseline characteristics. Contemp Clin Trials. 2024 Feb;137:107423. doi: 10.1016/j.cct.2023.107423. Epub 2023 Dec 25. PMID 38151173